CLINICAL TRIAL: NCT06001606
Title: Immunogenicity, Reactogenicity and Safety of 2 Doses of an Adjuvanted Herpes Zoster Subunit Vaccine in Patients With Systemic Lupus Erythematosus: a Randomized Clinical Trial.
Brief Title: Immunogenicity, Reactogenicity of Shingrix in SLE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-2303-017-1410
Record Dates: First submitted 2023-05-01; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-04

CONDITIONS: Zoster; Systemic Lupus Erythematosus; Vaccine Reaction
MeSH Terms: conditions — Herpes Zoster; Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shingrix (Experimental)
  Interventions: Drug: Shingrix
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Shingrix — Shingrix vaccination
  Arms: Shingrix
Drug: Placebo — Placebo vaccination
  Arms: Placebo

SUMMARY:
To investigate the immunogenicity, reactogenicity and safety of 2 doses of the adjuvanted herpes zoster subunit vaccine (Shingrix) in patients with SLE in a randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥ 19 years of age at time of consent
* ≥4 of the 1997 ACR13 or the 2012 SLICC/ACR criteria for SLE (13, 14)
* Clinically stable SLE
* Corticosteroid use: ≥ 5mg/day of prednisolone equivalent
* Stable dose of one or more of the following immunosuppressive treatment ≥ 4 weeks

  * Antimalarials (≤400 mg/day)
  * Azathioprine (≤3 mg/kg/day)
  * Mycophenolate mofetil (≤3 mg/day)
  * Tacrolimus (≤5mg/day)
  * Methotrexate (≤20mg/week)
  * Cyclosphosphamide (≤1mg/BSA/month)
* Must understand and voluntarily sign an informed consent form including writing consent for data protection

Exclusion Criteria:

* Pregnant or lactating females
* Acute infection with T >38°C at the time of vaccination
* Previous anaphylactic response to vaccine components or to egg
* History of Guillain-Barre syndrome or demyelinating syndromes
* Any condition including laboratory abnormality which places the subject at unacceptable risk
* Subjects who decline to participate

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2025-04-24 (Estimated); Study Completion 2025-04-24 (Estimated)

PRIMARY OUTCOMES:
Frequency of positive humoral vaccine response at 1 month post-dose 2 | 3 months
  Proporition of pariticpants who achieved a ≥4-fold increase in the anti-gE antibody concentration as compared to the prevaccination concentration

SECONDARY OUTCOMES:
Frequency of positive humoral vaccine response at 6 months post-dose 2 | 8 months
Frequency of humoral responses 12 month post-dose 2 | 14 month
Anti-gE antibody concentration at 6 months post-dose 2 | 8 months
Anti-gE antibody concentration at 12 months post-dose 2 | 14 months

OTHER OUTCOMES:
SLE flare rate | up to 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Park JK, Lee YJ, Shin K, Kang EH, Ha YJ, Park JW, Kim MJ, Kim MH, Choi SR, Jung Y, Lee JH, In Jung J, Kim JY, Winthrop KL, Lee EB. A Multicenter, Prospective, Randomized, Parallel-Group Trial on the Effects of Temporary Methotrexate Discontinuation for One Week Versus Two Weeks on Seasonal Influenza Vaccination in Patients With Rheumatoid Arthritis. Arthritis Rheumatol. 2023 Feb;75(2):171-177. doi: 10.1002/art.42318. Epub 2022 Dec 7. PMID 35930728
- [Result] Park JK, Lee MA, Lee EY, Song YW, Choi Y, Winthrop KL, Lee EB. Effect of methotrexate discontinuation on efficacy of seasonal influenza vaccination in patients with rheumatoid arthritis: a randomised clinical trial. Ann Rheum Dis. 2017 Sep;76(9):1559-1565. doi: 10.1136/annrheumdis-2017-211128. Epub 2017 May 3. PMID 28468794
- [Result] Park JK, Lee YJ, Shin K, Ha YJ, Lee EY, Song YW, Choi Y, Winthrop KL, Lee EB. Impact of temporary methotrexate discontinuation for 2 weeks on immunogenicity of seasonal influenza vaccination in patients with rheumatoid arthritis: a randomised clinical trial. Ann Rheum Dis. 2018 Jun;77(6):898-904. doi: 10.1136/annrheumdis-2018-213222. Epub 2018 Mar 23. PMID 29572291
- [Derived] Park JK, Kim M, Jung JI, Kim JY, Jeong H, Park JW, Winthrop KL, Lee EB. Immunogenicity, reactogenicity, and safety of two-dose adjuvanted herpes zoster subunit vaccine in patients with systemic lupus erythematosus in South Korea: a single-centre, randomised, double-blind, placebo-controlled trial. Lancet Rheumatol. 2024 Jun;6(6):e352-e360. doi: 10.1016/S2665-9913(24)00084-5. Epub 2024 May 3. PMID 38710192